CLINICAL TRIAL: NCT05871554
Title: Efficacy of a Brief Online Mindfulness and Self-Compassion Intervention (Mind-OP+) to Increase Connectedness: Randomized Controlled Trial
Brief Title: Efficacy of a Brief Online Mindfulness and Self-Compassion Intervention (Mind-OP+) to Increase Connectedness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-132
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Depression; Stress; Social Isolation; Anxiety
MeSH Terms: conditions — Depression; Social Isolation; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist (No Intervention): Participants are allocated to a waitlist condition where they participate in surveys for 11 weeks. Participants receive access to the treatment modules after completing the final survey after the 11th week.
- Treatment (Experimental): Participants are allocated to a treatment condition where they participate in surveys and online video modules for 11 weeks.
  Interventions: Behavioral: Mind-OP+

INTERVENTIONS:
Behavioral: Mind-OP+ — Mind-OP is an online program designed to cultivate mindfulness and self-compassion developed by Beshai and his team. Mind-OP is self-guided, with four modules administered at a pace of one module per week (four weeks total). The version used for this study, Mind-OP+, is five weeks total, containing an extra module focused on connectedness.
  The modules contain psychoeducational videos, guided audio meditations, goal-setting and motivational interviewing inspired exercises. Participants also have opportunities to engage with meditations and other exercises embedded within each module.
  The first module (Week 1) introduces the concept of mindfulness. The second module (Week 2) focuses on attention to bodily sensations and thoughts. The third module (Week 3) introduces the concept of self-compassion. The fourth module (Week 4) focuses on the self-kindness component of self-compassion. The fifth module (Week 5) focuses on the concept of connectedness.
  Arms: Treatment

SUMMARY:
Undergraduate students partook in an augmented, brief, online mindfulness and self-compassion-based program (Mind-OP+) to facilitate perceptions of connectedness. Participants were randomized into Mind-OP+ or waitlist control groups. It is hypothesized that connectedness at baseline will be negatively associated with mental health symptoms (depression, anxiety) and stress, and positively associated with self-compassion and dispositional mindfulness. Further, it is predicted that participants in the Mind-OP+ group will experience increases in connectedness compared with participants in the waitlist control condition. This study could provide support for a brief, convenient program to increase perceived connectedness, and thereby provide an option for students seeking protective factors for mental health and general resiliency.

DETAILED DESCRIPTION:
All measures, modules and questionnaires were hosted on Qualtrics, an online surveying software.

Upon signing up for the study and providing written informed consent, participants had access to a pre-treatment package via a Qualtrics link, which consisted of a consent form, demographic questions, and all measures (SCS-SF, FCS, FFMQ-15, SNI, RNS, SCS-R, and DASS-21). Within one week of participants completing the pre-treatment package, the principal investigator sorted through the data to determine eligibility based on symptom criteria (mild to moderate depression and/or anxiety symptoms, and/or mild to moderate stress levels). Those who met criteria were randomly assigned to the waitlist group or treatment group using Research Randomizer, a web-based pseudo-random number generator. The principal investigator e-mailed ineligible participants, thanked them for their time, as well as provided them with a debriefing form and links to the Mind-OP+ modules for their personal use.

Each week for five weeks, the treatment group was emailed a package containing the Mind-OP+ module, the symptom measure (DASS-21), and the connectedness measures (SCS-R, RNS, and SNI). Additionally, other outcome measures (SCS-SF, FCS, and FFMQ-15) were e-mailed in the middle of the trial at the three-week point. The waitlist group received an e-mail with a Qualtrics link containing the same measures following the same schedule, but without the Mind-OP+ modules. The principal investigator sent reminders twice a week to both groups to ensure that participants were completing the packages, as a previous student trial of Mind-OP following the same reminder schedule had 59% of enrolled participants complete the intervention (Bueno et al., in preparation).

After completion of the five-week intervention, on the seventh week of the trial, all participants received the post-treatment package that contains all measures (SCS-SF, FCS, FFMQ-15, SNI, RNS, SCS-R, and DASS-21. One month following the completion of the study, all participants received another follow-up package containing all measures, a debrief form, and access to mental health resources. At this point, the principal investigator e-mailed the intervention modules to the waitlist group.

Following completion of data collection, the principal investigator conducted ten correlation analyses to examine zero-order correlation coefficients of baseline SCS-R and RNS scores with baseline DASS-21, FFMQ-15, FCS, SCS-SF, and SCS-SF - Common Humanity Subscale (SCS-SF-CH) scores. Two multilevel modeling analyses (MLM) were conducted to compare changes in scores on relatedness and social connectedness between the treatment group (Mind-OP+) and waitlist group over the 12-week trial duration (7-week intervention duration + at the one-month follow-up). Four serial mediation models analysed whether changes in mindfulness and self-compassion mediated relationships between treatment outcomes for both groups and changes in relatedness and social connectedness. Further, SNI scores were examined using two exploratory sign tests.

ELIGIBILITY:
Inclusion Criteria:

* University student
* Mild to moderate levels of anxiety, depression, and/or stress

Exclusion Criteria:

* Non university students
* Below mild levels of anxiety, depression, and stress

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Relatedness Needs Subscale (RNS) | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, and Week 11
  Change from Baseline in Relatedness Scores at Weeks 1-6 and Week 11. Total score range: 1-7. Lower values are indicative of lower relatedness needs satisfaction (a worse outcome). Total scores are computed by summing all scale items and calculating an average.
The Social Connectedness Scale - Revised (SCS-R) | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, and Week 11
  Change from Baseline in Social Connectedness Scores at Weeks 1-6 and Week 11. Total score range: 20 - 120. Lower values are indicative of lower levels of social connectedness (a worse outcome). Total scores are computed by summing all scale items.
Berkman-Syme Social Network Index (SNI) | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, and Week 11
  Change from Baseline in Social Network Scores at Weeks 1-6 and Week 11. Total score range: 0-4. Lower scores are indicative of more isolation (a worse outcome). Total score is a composite score calculated by assigning one point for each relationship category endorsed (i.e., marriage, friends, relatives, and group activities) for up to a total of 4 points.

SECONDARY OUTCOMES:
The Depression, Anxiety, and Stress Scale - 21 Items (DASS-21) | Baseline, Week 6, and Week 11
  Change from Baseline in Depression, Anxiety and Stress Scores at Week 6 and Week 11. Total score range: 0 - 126. Lower scores are indicative of less symptoms of depression and anxiety and lower levels of stress (a better outcome). Total score is calculated by summing scale items and multiplying by 2.
The Five-Facet Mindfulness Questionnaire 15 (FFMQ-15) | Baseline, Week 6, and Week 11
  Change from Baseline in Mindfulness Scores at Week 6 and Week 11. Total score range: 15 - 75. Lower scores are indicative of less trait mindfulness (worse outcome). Total score is computed by summing all scale items.
Fears of Compassion Scale (FCS) | Baseline, Week 6, and Week 11
  Change from Baseline in Fears of Compassion Scores at Week 6 and Week 11. Total score range: 0 - 152. Lower scores are indicative of less fears of compassion (better outcome). Total score is computed by summing all scale items.
The Self-Compassion Scale-Short Form (SCS-SF) | Baseline, Week 6, and Week 11
  Change from Baseline in Self-Compassion Scores at Week 6 and Week 11. Total score range: 1 - 5. Lower scores are indicative of less self-compassion (worse outcome). Total score is computed by summing all items and calculating an average.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Bueno, B.A. (Hons), Principal Investigator — University of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

REFERENCES:
- [Background] Beshai S, Bueno C, Yu M, Feeney JR, Pitariu A. Examining the effectiveness of an online program to cultivate mindfulness and self-compassion skills (Mind-OP): Randomized controlled trial on Amazon's Mechanical Turk. Behav Res Ther. 2020 Nov;134:103724. doi: 10.1016/j.brat.2020.103724. Epub 2020 Sep 10. PMID 32942203